CLINICAL TRIAL: NCT04168294
Title: The Influence of Sedation for Endoscopy on Cognitive Function
Status: Terminated | Type: Observational
Why Stopped: The number of subjects did not meet the requirements
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Ren Ji Hospital, School of medicine, Shanghai Jiao Tong University, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjyyxhk2017001
Record Dates: First submitted 2018-09-26; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Esophagogastroduodenoscopy; Deep Sedation; Cognition Disorders
Keywords: Esophagogastroduodenoscopy; Deep Sedation; Cognition Disorders; Patient Discharge; Automobile Driving
MeSH Terms: conditions — Cognition Disorders | interventions — Propofol; Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- sedation group: Patients undergo sedative esophagogastroduodenoscopy (EGD) and are intravenous injected propofol in bolus
  Interventions: Drug: Propofol; Device: endoscopy
- control group: patients undergo conventional EGD
  Interventions: Device: endoscopy

INTERVENTIONS:
Drug: Propofol — patients in sedation group will be intravenous injected propofol in bolus
  Groups: sedation group
Device: endoscopy — endoscopy system
  Other Names: Olympus Lucera Elite 290 system

SUMMARY:
It is commonly recommended that patients should refrain from driving for 24 hours after sedation for endoscopy，however，this recommendation has been queried recently．To investigate the effect of sedation on early postoperative cognitive function in patients undergoing endoscopy.

DETAILED DESCRIPTION:
One hundred adult patients undergoing sedative esophagogastroduodenoscopy ( EGD) were randomly recruited，and another 100 adult patients undergoing conventional（without sedation） EGD were served as controls． All patients had an education level more than 9 years． Cognitive function was assessed by Montreal Cognitive Assessment（MoCA）1 week before EGD exam, 10 mins before propofol sedation or the beginning of endoscopic procedure, 30mins after EGD exam, and 2 week after exam.

ELIGIBILITY:
Inclusion Criteria:

1. The scores of MMSE are more than 26.
2. The AHA grade I and II.

Exclusion Criteria:

1. The AHA grade III, IV or V.
2. binge drinking.
3. Take sedatives, sleeping agents and some drug which may affect the study in a month.
4. Psychiatric disorders.
5. The dysfunction of heart, lung, liver and kidney.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Radom select patients who undergo EGD in Renji Hospital, School of Medicine, Shanghai Jiaotong University. Patients who are recruited all received nine year compulsory education and fit for the inclusion criteria. Moreover, all patients received approval from the local institutional review board.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
NCT-A test outcome measure | 30 minutes
  the score of NCT-A test for each patient is not less than that in the baseline.
DST test outcome measure | 30 minutes
  the score of DST for each patient is not less than that in the baseline.
number cancellation test outcome measure | 30 minutes
  the score of number cancellation test for each patient is not less than that in the baseline.

SECONDARY OUTCOMES:
heart rate outcome measure | 5 minutes
  heart rate less than 50 time per minute
SpO2 outcome measure | 5 minutes
  SpO2 less than 90%

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Ping Li, Study Chair — Renji Hospital, School of Medicine,Shanghai Jiao Tong University
Locations (1):
- Department of Gastroenterology, Renji Hospital, Shanghai Institute of Digestive Diseases, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided